CLINICAL TRIAL: NCT00468650
Title: A Multicenter, Open Label, High Dose (100mg) Rapid Titration Study, To Evaluate The Efficacy And Satisfaction Of Patrex® (Sildenafil Citrate) In Men With Erectile Dysfunction In Mexico.
Brief Title: A Multicenter, Open Label, To Evaluate The Efficacy And Satisfaction Of Patrex® In Men With Erectile Dysfunction.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1481251
Record Dates: First submitted 2007-05-01; First posted 2007-05-03 (Estimated); Results first posted 2009-03-16 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Active Comparator): Eligible patients fulfilling all inclusion/exclusion criteria will be assigned at Visit 2/Week 0 (Baseline) to receive Patrex® 50 mg as needed (PRN) during the first two weeks, and,thereafter, at Visit 3/Week 2, all enrolled subjects will be up titrated to Patrex® 100 mg PRN for the following four weeks.
  Interventions: Drug: sildenafil citrate

INTERVENTIONS:
Drug: sildenafil citrate — Tablets, 50mg and 100mg , Medication will be taken orally with a glass of water approximately one hour (30 min to 4 hours) before sexual activity. Subjects are to take one dose in any calendar day.Eligible patients fulfilling all inclusion/exclusion criteria will be assigned at Visit 2/Week 0 (Baseline) to receive sildenafil 50 mg as needed (PRN) during the first two weeks, and,thereafter, at Visit 3/Week 2, all enrolled subjects will be up titrated to sildenafil 100 mg PRN for the following four weeks.

SUMMARY:
A multicenter open label study to assess the efficacy of sildenafil rapid dose titration to 100 mg in men with erectile dysfunction, based on the Erectile Function (EF) domain score of the International Index of Erectile Function (IIEF) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Documented Clinical diagnosis of Erectile Dysfunction (ED) by International Index of Erectile Function (IIEF) Erectile Function (EF) Domain score less than or equal to 25.
* Subjects must be in a stable relationship

Exclusion Criteria:

* Subject with resting sitting hypotension (BP <90/50 mmHg) or hypertension (BP>170/110 mmHg) and orthostatic hypotension.
* Subjects receiving any PDE (Phosphodiesterase)-5 inhibitors within 4 weeks prior to the date of screening.
* Subjects with severe hepatic impairment, a known history of retinitis pigmentare.
* Subjects with significant cardiovascular disease in the last 3 months (per medical history.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Mexico (7):
  - Pfizer Investigational Site, México, D.F.
  - Pfizer Investigational Site, Naucalpan, Edo. de México
  - Pfizer Investigational Site, Zapopan, Jalisco
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Aguascalientes
  - Pfizer Investigational Site, Durango
  - Pfizer Investigational Site, Naucalpan Edo. de Mexico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481251&StudyName=A%20Multicenter%2C%20Open%20Label%2C%20%20To%20Evaluate%20The%20Efficacy%20And%20Satisfaction%20Of%20Patrex%AE%20In%20Men%20With%20Erectile%20Dysfunction.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible subjects had to have at least 2 attempts at sexual intercourse during the 2 week screening phase to begin the sildenafil citrate 50mg treatment at baseline.
Groups:
- Open Label Sildenafil Citrate: Eligible patients fulfilling all inclusion/exclusion criteria will be assigned at Visit 2/Week 0 (Baseline) to receive sildenafil citrate 50 mg as needed (PRN) during the first two weeks, and,thereafter, at Visit 3/Week 2, all enrolled subjects will be up titrated to sildenafil citrate 100 mg PRN for the following four weeks.
Period: Overall Study
Arm/Group | Open Label Sildenafil Citrate
Started | 117
Completed | 110
Not Completed | 7
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 117

OUTCOME MEASURES:

1. Primary Outcome: International Index of Erectile Function (IIEF), Erectile Function (EF) Domain Score- Change From Baseline to Week 6 Last Observation Carried Forward (LOCF)
Description: IIEF is a self-administered scale designed to assess erectile functioning: includes 15 questions on 5 relevant domains of male sexual function; one is erectile function (EF). IIEF-EF Domain: sum of scores for Questions 1, 2, 3, 4, 5 & 15 from IIEF. Score range: 0 to 5 (Q1 to Q5), 1 to 5 (Q15); total 1 to 30. Higher score indicates better outcome.
Time Frame: Week 6 LOCF
Population: Modified intent to treat (MITT) population consists of subjects in the safety population who provided at least 1 post baseline efficacy assessment. The Week 6 Last Observation Carried Forward (LOCF) value is the last post-baseline value, ie, last assessment collected at visits after Visit 1. Week 6 Endpoint = last observation recorded after Week 2.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 113
score on scale | 10.96 (5.19)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Primary hypothesis to be tested is whether there is a significant improvement in the IIEF EF domain at the end of the 100 mg period, as compared to the baseline (Week 0) score. Sample size (N=115) provides more than 90% power to detect a change from baseline of 10 in the primary efficacy variable, assuming a standard deviation of 9, using the two-sided, single-sample t-test with significance level (alpha) of 0.05; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Statistical significance will be declared if the p-value is <0.05. Change from Baseline: Week 6 (LOCF) minus Baseline; single sample t-test; Mean Difference (Net) = 10.96, 95% CI [10.00 to 11.93], Standard Deviation 5.19

2. Secondary Outcome: International Index of Erectile Function (IIEF), Erectile Function (EF) Domain Score - Change From Baseline at Weeks 2, 4 and 6
Description: as for outcome 1
Time Frame: Week 2, Week 4 and Week 6
Population: MITT population consists of subjects in the safety population who provided at least 1 post baseline efficacy assessment. Week 6 Endpoint = last observation recorded after Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 113
score on a scale
  Week 2 (N=113) | 7.14 (5.21)
  Week 4 (N=112) | 10.57 (5.43)
  Week 6 (N=110) | 10.93 (5.26)
  Week 6 Endpoint (N=112) | 10.95 (5.21)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 7.14, 95% CI [6.17 to 8.11], Standard Deviation 5.21
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 10.57, 95% CI [9.56 to 11.59], Standard Deviation 5.43
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 10.93, 95% CI [9.93 to 11.92], Standard Deviation 5.26
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 endpoint minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 10.95, 95% CI [9.97 to 11.92], Standard Deviation 5.21

3. Secondary Outcome: International Index of Erectile Function (IIEF), Erectile Function (EF) Domain Score- Change From Week 2
Description: as for outcome 1
Time Frame: Week 4 and Week 6
Population: MITT population consists of subjects in the safety population who provided at least 1 post baseline efficacy assessment. The Week 6 Last Observation Carried Forward (LOCF) value is the last post-baseline value, ie, the last assessment among those collected at visits after Visit 1. Week 6 Endpoint = last observation recorded after Week 2
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Open Label Sildenafil Citrate: Eligible patients fulfilling all inclusion/exclusion criteria will be assigned at Visit 2/Week 0 (Baseline) to receive sildenafil citrate 50 mg as needed (PRN) during the first two weeks, and, thereafter, at Visit 3/Week 2, all enrolled subjects will be up titrated to sildenafil citrate 100 mg PRN for the following four weeks.
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
score on scale
  Week 4 (N=112) | 3.48 (3.97)
  Week 6 (N=110) | 3.88 (4.38)
  Week 6 LOCF (N=112) | 3.86 (4.35)
  Week 6 Endpoint (N=112) | 3.86 (4.35)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.48, 95% CI [2.74 to 4.23], Standard Deviation 3.97
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2 For the secondary outcome, the change in IIEF-EF domain from the end of 50 mg period (Week 2) to the end of 100 mg period (Week 6), the sample size (N=115) provides more than 80% power to detect a mean change of 1.75 points, assuming a standard deviation of 6, using the two-sided, single sample t-test with significance level (alpha) of 0.05; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.88, 95% CI [3.05 to 4.71], Standard Deviation 4.38
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2 For the secondary outcome, the change in IIEF-EF domain from the end of 50 mg period (Week 2) to the end of 100 mg period (Week 6), the sample size (N=115) provides more than 80% power to detect a mean change of 1.75 points, assuming a standard deviation of 6, using the two-sided, single sample t-test with significance level (alpha) of 0.05; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.86, 95% CI [3.04 to 4.67], Standard Deviation 4.35
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2 For the secondary outcome, the change in IIEF-EF domain from the end of 50 mg period (Week 2) to the end of 100 mg period (Week 6), the sample size (N=115) provides more than 80% power to detect a mean change of 1.75 points, assuming a standard deviation of 6, using the two-sided, single sample t-test with significance level (alpha) of 0.05; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.86, 95% CI [3.04 to 4.67], Standard Deviation 4.35

4. Secondary Outcome: International Index of Erectile Function (IIEF), Orgasmic Function Domain- Change From Baseline
Description: IIEF is a self-administered scale to assess erectile functioning. IIEF includes 15 questions and addresses the 5 relevant domains of male sexual function, one is orgasmic function. IIEF Orgasmic Function Domain was sum of scores for Questions 9 and 10 from the IIEF. Score range: 0 to 5; total 0 to 10. Higher score indicates better outcome.
Time Frame: Week 2, Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 113
score on scale
  Week 2 (N=113) | 1.89 (2.40)
  Week 4 (N=112) | 2.46 (2.32)
  Week 6 (N=110) | 2.59 (2.44)
  Week 6 LOCF (N=113) | 2.63 (2.45)
  Week 6 Endpoint (N=112) | 2.59 (2.42)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for significance p<0.05; single sample t-test; Mean Difference (Net) = 1.89, 95% CI [1.45 to 2.34], Standard Deviation 2.40
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 2.46, 95% CI [2.02 to 2.89], Standard Deviation 2.32
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 2.59, 95% CI [2.13 to 3.05], Standard Deviation 2.44
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 2.63, 95% CI [2.17 to 3.08], Standard Deviation 2.45
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 2.59, 95% CI [2.14 to 3.04], Standard Deviation 2.42

5. Secondary Outcome: International Index of Erectile Function (IIEF), Orgasmic Function Domain- Change From Week 2
Description: as for outcome 4
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
score on scale
  Week 4 (N=112) | 0.61 (1.51)
  Week 6 (N=110) | 0.75 (1.46)
  Week 6 LOCF (N=112) | 0.74 (1.45)
  Week 6 Endpoint (N=112) | 0.74 (1.45)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 0.61, 95% CI [0.32 to 0.89], Standard Deviation 1.51
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 0.75, 95% CI [0.47 to 1.02], Standard Deviation 1.46
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 0.74, 95% CI [0.47 to 1.01], Standard Deviation 1.45
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 0.74, 95% CI [0.47 to 1.01], Standard Deviation 1.45

6. Secondary Outcome: International Index of Erectile Function (IIEF), Sexual Desire Domain Score- Change From Baseline
Description: IIEF is a self-administered scale to assess erectile functioning. IIEF includes 15 questions and addresses the 5 relevant domains of male sexual function, one of which is sexual desire. IIEF Sexual Desire Domain was sum of scores for Questions 11 and 12 from the IIEF. Score range: 1 to 5; total 2 to 10. Higher score indicates better outcome.
Time Frame: Week 2, Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 113
score on scale
  Week 2 (N=113) | 1.43 (1.87)
  Week 4 (N=112) | 2.00 (1.86)
  Week 6 (N=110) | 2.25 (1.91)
  Week 6 LOCF (N=113) | 2.26 (1.94)
  Week 6 Endpoint (N=112) | 2.28 (1.93)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.43, 95% CI [1.09 to 1.78], Standard Deviation 1.87
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 2.00, 95% CI [1.65 to 2.35], Standard Deviation 1.86
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 2.25, 95% CI [1.89 to 2.62], Standard Deviation 1.91
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 2.26, 95% CI [1.90 to 2.62], Standard Deviation 1.94
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 2.28, 95% CI [1.91 to 2.64], Standard Deviation 1.93

7. Secondary Outcome: International Index of Erectile Function (IIEF), Sexual Desire Domain Score- Change From Week 2
Description: as for outcome 6
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
score on scale
  Week 4 (N=112) | 0.55 (1.41)
  Week 6 (N=110) | 0.81 (1.47)
  Week 6 LOCF (N=112) | 0.83 (1.49)
  Week 6 Endpoint (N=112) | 0.83 (1.49)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 0.55, 95% CI [0.29 to 0.82], Standard Deviation 1.41
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 0.81, 95% CI [0.53 to 1.09], Standard Deviation 1.47
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 0.83, 95% CI [0.55 to 1.11], Standard Deviation 1.49
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 0.83, 95% CI [0.55 to 1.11], Standard Deviation 1.49

8. Secondary Outcome: International Index of Erectile Function (IIEF), Intercourse Satisfaction Domain Score- Change From Baseline
Description: IIEF is a self-administered scale to assess erectile functioning. IIEF includes 15 questions and addresses the 5 relevant domains of male sexual function, one is intercourse satisfaction. IIEF Intercourse Satisfaction Domain: sum of scores for Questions 6, 7 and 8 from IIEF. Score range: 0 to 5; total 0 to 15. Higher score indicates better outcome.
Time Frame: Week 2, Week 4, and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 113
score on scale
  Week 2 (N=113) | 3.18 (2.42)
  Week 4 (N=112) | 4.38 (2.39)
  Week 6 (N=110) | 4.73 (2.53)
  Week 6 LOCF (N=113) | 4.70 (2.52)
  Week 6 Endpoint (N=112) | 4.72 (2.52)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.18, 95% CI [2.73 to 3.63], Standard Deviation 2.42
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 4.38, 95% CI [3.94 to 4.83], Standard Deviation 2.39
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 4.73, 95% CI [4.25 to 5.21], Standard Deviation 2.53
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 4.70, 95% CI [4.23 to 5.17], Standard Deviation 2.52
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 4.72, 95% CI [4.25 to 5.19], Standard Deviation 2.52

9. Secondary Outcome: International Index of Erectile Function (IIEF), Intercourse Satisfaction Domain Score- Change From Week 2
Description: as for outcome 8
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
score on scale
  Week 4 (N=112) | 1.20 (2.10)
  Week 6 (N=110) | 1.54 (2.20)
  Week 6 LOCF (N=112) | 1.54 (2.19)
  Week 6 Endpoint (N=112) | 1.54 (2.19)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.20, 95% CI [0.80 to 1.59], Standard Deviation 2.10
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.54, 95% CI [1.12 to 1.95], Standard Deviation 2.20
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.54, 95% CI [1.13 to 1.95], Standard Deviation 2.19
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.54, 95% CI [1.13 to 1.95], Standard Deviation 2.19

10. Secondary Outcome: International Index of Erectile Function (IIEF), Overall Satisfaction Domain Score- Change From Baseline
Description: IIEF is a self-administered scale to assess erectile functioning. IIEF includes 15 questions and addresses the 5 relevant domains of male sexual function, one is overall satisfaction. IIEF Overall Satisfaction Domain was sum of scores for Questions 13 and 14 from the IIEF. Score range: 1 to 5; total 2 to 10. Higher score indicates better outcome.
Time Frame: Week 2, Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 113
score on scale
  Week 2 (N=113) | 2.73 (2.38)
  Week 4 (N=112) | 3.67 (2.49)
  Week 6 (N=110) | 3.92 (2.52)
  Week 6 LOCF (N=113) | 3.91 (2.53)
  Week 6 Endpoint (N=112) | 3.89 (2.53)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 2.73, 95% CI [2.28 to 3.17], Standard Deviation 2.38
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.67, 95% CI [3.20 to 4.14], Standard Deviation 2.49
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.92, 95% CI [3.44 to 4.40], Standard Deviation 2.52
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.91, 95% CI [3.44 to 4.38], Standard Deviation 2.53
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.89, 95% CI [3.42 to 4.37], Standard Deviation 2.53

11. Secondary Outcome: International Index of Erectile Function (IIEF), Overall Satisfaction Domain Score- Change From Week 2
Description: as for outcome 10
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
score on scale
  Week 4 (N=112) | 0.97 (1.88)
  Week 6 (N=110) | 1.21 (1.92)
  Week 6 LOCF (N=112) | 1.20 (1.90)
  Week 6 Endpoint (N=112) | 1.20 (1.90)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 0.97, 95% CI [0.62 to 1.32], Standard Deviation 1.88
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.21, 95% CI [0.85 to 1.57], Standard Deviation 1.92
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.20, 95% CI [0.84 to 1.55], Standard Deviation 1.90
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.20, 95% CI [0.84 to 1.55], Standard Deviation 1.90

12. Secondary Outcome: Quality of Erection Questionnaire (QEQ): Total Score - Change From Baseline
Description: QEQ is a self-administered scale used to assess erection hardness and overall quality of erections. The QEQ total score is defined as the sum of the scores from QEQ Questions 1-6. Score range: 1 to 5. Higher score indicates better outcome. Raw QEQ score ranges from 6-30 and is transformed onto a 0-100 scale.
Time Frame: Week 2, Week 4, and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 113
score on scale
  Week 2 (N=113) | 32.71 (25.36)
  Week 4 (N=112) | 46.21 (26.27)
  Week 6 (N=110) | 45.53 (26.96)
  Week 6 LOCF (N=113) | 45.28 (27.01)
  Week 6 Endpoint (N=112) | 45.05 (27.02)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 32.71, 95% CI [27.98 to 37.43], Standard Deviation 25.36
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 46.21, 95% CI [41.29 to 51.12], Standard Deviation 26.27
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 45.53, 95% CI [40.44 to 50.63], Standard Deviation 26.96
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 45.28, 95% CI [40.25 to 50.31], Standard Deviation 27.01
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 45.05, 95% CI [39.99 to 50.11], Standard Deviation 27.02

13. Secondary Outcome: Quality of Erection Questionnaire (QEQ): Total Score- Change From Week 2
Description: as for outcome 12
Time Frame: Week 4 and Week 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 113
score on scale
  Week 4 (N=112) | 13.84 (21.10)
  Week 6 (N=110) | 13.07 (24.25)
  Week 6 LOCF (N=112) | 12.69 (24.26)
  Week 6 Endpoint (N=112) | 12.69 (24.26)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 13.84, 95% CI [9.89 to 17.79], Standard Deviation 21.10
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 13.07, 95% CI [8.49 to 17.65], Standard Deviation 24.25
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 12.69, 95% CI [8.14 to 17.23], Standard Deviation 24.26
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 12.69, 95% CI [8.14 to 17.23], Standard Deviation 24.26

14. Secondary Outcome: Sexual Experience Questionnaire (Sex-Q): Erection Domain - Change From Baseline
Description: Sexual Experience Questionnaire (Sex-Q) is a self-administered questionnaire designed to assess functional, emotional, and social aspects of sexual experience. Sex-Q includes 15 questions. Sex-Q Erection domain: sum of scores for Questions 1, 2, 3, 4, 5 and 6 from the Sex-Q. Score range: 1 to 5; total 6 to 30. Higher score indicates better outcome.
Time Frame: Week 2, Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 113
score on scale
  Week 2 (N=113) | 5.41 (4.40)
  Week 4 (N=112) | 8.85 (4.96)
  Week 6 (N=110) | 9.21 (5.19)
  Week 6 LOCF (N=113) | 9.28 (5.14)
  Week 6 Endpoint (N=112) | 9.25 (5.15)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 5.41, 95% CI [4.59 to 6.23], Standard Deviation 4.40
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 8.85, 95% CI [7.92 to 9.78], Standard Deviation 4.96
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 9.21, 95% CI [8.23 to 10.19], Standard Deviation 5.19
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 9.28, 95% CI [8.32 to 10.24], Standard Deviation 5.14
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 9.25, 95% CI [8.28 to 10.22], Standard Deviation 5.15

15. Secondary Outcome: Sexual Experience Questionnaire (Sex-Q): Erection Domain- Change From Week 2
Description: as for outcome 14
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
score on scale
  Week 4 (N=112) | 3.51 (3.89)
  Week 6 (N=110) | 3.91 (4.41)
  Week 6 LOCF (N=112) | 3.91 (4.38)
  Week 6 Endpoint (N=112) | 3.91 (4.38)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.51, 95% CI [2.78 to 4.24], Standard Deviation 3.89
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.91, 95% CI [3.08 to 4.74], Standard Deviation 4.41
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.91, 95% CI [3.09 to 4.73], Standard Deviation 4.38
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.91, 95% CI [3.09 to 4.73], Standard Deviation 4.38

16. Secondary Outcome: Sexual Experience Questionnaire (Sex-Q): Satisfaction Domain - Change From Baseline
Description: Sexual Experience Questionnaire (Sex-Q) is a self-administered questionnaire designed to assess functional, emotional, and social aspects of sexual experience. Sex-Q includes 15 questions (q). Sex-Q Satisfaction domain:sum of scores for q 10, 11, 12, 13, 14 and 15 from Sex-Q. Score range:1 to 5; total 6 to 30. Higher score indicates better outcome
Time Frame: Week 2, Week 4, and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 113
score on scale
  Week 2 (N=113) | 6.68 (4.86)
  Week 4 (N=112) | 9.94 (5.21)
  Week 6 (N=108) | 10.59 (5.08)
  Week 6 LOCF (N=111) | 10.63 (5.03)
  Week 6 Endpoint (N=110) | 10.64 (5.06)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 6.68, 95% CI [5.77 to 7.59], Standard Deviation 4.86
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 9.94, 95% CI [8.96 to 10.91], Standard Deviation 5.21
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 10.59, 95% CI [9.62 to 11.56], Standard Deviation 5.08
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 10.63, 95% CI [9.68 to 11.58], Standard Deviation 5.03
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 10.64, 95% CI [9.68 to 11.59], Standard Deviation 5.06

17. Secondary Outcome: Sexual Experience Questionnaire (Sex-Q): Satisfaction Domain - Change From Week 2
Description: as for outcome 16
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
score on scale
  Week 4 (N=112) | 3.29 (4.10)
  Week 6 (N=108) | 4.03 (5.09)
  Week 6 LOCF (N=110) | 4.01 (5.04)
  Week 6 Endpoint (N=110) | 4.01 (5.04)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.29, 95% CI [2.52 to 4.05], Standard Deviation 4.10
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 4.03, 95% CI [3.06 to 5.00], Standard Deviation 5.09
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 4.01, 95% CI [3.06 to 4.96], Standard Deviation 5.04
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 4.01, 95% CI [3.06 to 4.96], Standard Deviation 5.04

18. Secondary Outcome: Sexual Experience Questionnaire (Sex-Q): Relationship Domain - Change From Baseline
Description: Sexual Experience Questionnaire (Sex-Q) is a self-administered questionnaire designed to assess functional, emotional, and social aspects of sexual experience. Sex-Q includes 15 questions. Sex-Q Relationship domain was sum of scores for Questions 7, 8 and 9 from the Sex-Q. Score range: 1 to 5; total 3 to 15. Higher score indicates better outcome.
Time Frame: Week 2, Week 4, and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
score on scale
  Week 2 (N=112) | 2.79 (2.44)
  Week 4 (N=111) | 4.23 (2.56)
  Week 6 (N=108) | 4.74 (2.84)
  Week 6 LOCF (N=111) | 4.78 (2.81)
  Week 6 Endpoint (N=110) | 4.76 (2.82)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 2.79, 95% CI [2.33 to 3.24], Standard Deviation 2.44
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 4.23, 95% CI [3.74 to 4.71], Standard Deviation 2.56
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 4.74, 95% CI [4.20 to 5.28], Standard Deviation 2.84
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 4.78, 95% CI [4.25 to 5.31], Standard Deviation 2.81
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 4.76, 95% CI [4.23 to 5.30], Standard Deviation 2.82

19. Secondary Outcome: Sexual Experience Questionnaire (Sex-Q): Relationship Domain - Change From Week 2
Description: as for outcome 18
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
score on scale
  Week 4 (N=112) | 1.49 (1.91)
  Week 6 (N=109) | 1.96 (2.08)
  Week 6 LOCF (N=111) | 1.98 (2.07)
  Week 6 Endpoint (N=111) | 1.98 (2.07)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.49, 95% CI [1.13 to 1.85], Standard Deviation 1.91
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.96, 95% CI [1.57 to 2.36], Standard Deviation 2.08
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.98, 95% CI [1.59 to 2.37], Standard Deviation 2.07
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.98, 95% CI [1.59 to 2.37], Standard Deviation 2.07

20. Secondary Outcome: Mean Per-Patient Percentage of 'Yes' Responses to Sexual Encounter Profile (SEP) Question 1 on Occasions With Sexual Stimulation- Change From Baseline
Description: Mean change: mean change at each visit minus mean at baseline. Percent of "Yes" responses to Question 1 based on occasions (= sexual stimulation): 100*(number of occasions where SEP Question 1 [Were you able to achieve at least some erection (some enlargement of the penis)?] = Yes) / (number of occasions where Question 1 was answered Yes or No)
Time Frame: Week 2, Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 110
per-patient percentage
  Question 1 (Week 2) N=110 | 8.84 (28.70)
  Question 1 (Week 4) N=108 | 10.18 (27.51)
  Question 1 (Week 6) N=105 | 12.29 (28.88)
  Question 1 (Week 6 LOCF) N=110 | 11.96 (28.33)
  Question 1 (Week 6 Endpoint) N=108 | 11.95 (28.55)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus baseline; Test type: Superiority or Other; p = 0.0016, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Median Difference (Net) = 8.84, 95% CI [3.42 to 14.26], Standard Deviation 28.70
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 10.18, 95% CI [4.93 to 15.43], Standard Deviation 27.51
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 12.29, 95% CI [6.70 to 17.88], Standard Deviation 28.88
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 11.96, 95% CI [6.61 to 17.32], Standard Deviation 28.33
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 11.95, 95% CI [6.51 to 17.40], Standard Deviation 28.55

21. Secondary Outcome: Mean Per-Patient Percentage of 'Yes' Responses to Sexual Encounter Profile (SEP) Question 1 Based on Occasions With Sexual Stimulation- Change From Week 2
Description: Mean change: mean change at each visit minus mean at Week 2. Percent of "Yes" responses to Question 1 based on occasions (= sexual stimulation): 100*(number of occasions where SEP Question 1 [Were you able to achieve at least some erection (some enlargement of the penis)?] = Yes) / (number of occasions where Question 1 was answered Yes or No)
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 113
per-patient percentage
  Question 1 (Week 4) N=111 | 1.37 (14.85)
  Question 1 (Week 6) N=108 | 3.12 (14.26)
  Question 1 (Week 6 LOCF) N=113 | 2.98 (13.95)
  Question 1 (Week 6 Endpoint) N=111 | 3.04 (14.07)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p = 0.3324, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.37, 95% CI [-1.42 to 4.17], Standard Deviation 14.85
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p = 0.0249, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.12, 95% CI [0.40 to 5.84], Standard Deviation 14.26
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p = 0.0249, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 2.98, 95% CI [0.37 to 5.58], Standard Deviation 13.95
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p = 0.0249, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 3.04, 95% CI [0.39 to 5.68], Standard Deviation 14.07

22. Secondary Outcome: Mean Per-Patient Percentage of 'Yes' Responses to Sexual Encounter Profile (SEP) Question 2 on Occasions With Sexual Stimulation- Change From Baseline
Description: Mean change: mean change at each visit minus mean at baseline. Percent of "Yes" responses to SEP Question 2 based on occasions (= sexual stimulation): 100*(number of occasions where SEP Question 2 ["Were you able to insert your penis into your partner's vagina?"] = "Yes") / (number of occasions where SEP Question 2 was answered "Yes" or "No").
Time Frame: Week 2, Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 102
per-patient percentage
  Question 2 (Week 2) N=102 | 15.37 (30.51)
  Question 2 (Week 4) N=100 | 17.15 (32.22)
  Question 2 (Week 6) N=97 | 18.22 (32.44)
  Question 2 (Week 6 LOCF) N=102 | 17.33 (31.87)
  Question 2 (Week 6 Endpoint) N=100 | 17.68 (32.10)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 15.37, 95% CI [9.38 to 21.36], Standard Deviation 30.51
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 17.15, 95% CI [10.76 to 23.55], Standard Deviation 32.22
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 18.22, 95% CI [11.68 to 24.76], Standard Deviation 32.44
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 17.33, 95% CI [11.07 to 23.59], Standard Deviation 31.87
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 17.68, 95% CI [11.31 to 24.04], Standard Deviation 32.10

23. Secondary Outcome: Mean Per-Patient Percentage of 'Yes' Responses to Sexual Encounter Profile (SEP) Question 2 on Occasions With Sexual Stimulation- Change From Week 2
Description: Mean change: mean change at each visit minus mean at Week 2. Percent of "Yes" responses to SEP Question 2 based on occasions (= sexual stimulation): 100*(number of occasions where SEP Question 2 ["Were you able to insert your penis into your partner's vagina?"] = "Yes") / (number of occasions where SEP Question 2 was answered "Yes" or "No").
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
per-patient percentage
  Question 2 (Week 4) N=110 | 1.46 (9.41)
  Question 2 (Week 6) N=107 | 1.18 (12.33)
  Question 2 (Week 6 LOCF) N=112 | 1.13 (12.05)
  Question 2 (Week 6 Endpoint) N=110 | 1.15 (12.16)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p = 0.1061, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.46, 95% CI [-0.32 to 3.24], Standard Deviation 9.41
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p = 0.3237, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.18, 95% CI [-1.18 to 3.54], Standard Deviation 12.33
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p = 0.3236, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.13, 95% CI [-1.13 to 3.38], Standard Deviation 12.05
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p = 0.3236, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 1.15, 95% CI [-1.15 to 3.45], Standard Deviation 12.16

24. Secondary Outcome: Mean Per-Patient Percentage of 'Yes' Responses to Sexual Encounter Profile (SEP) Question 3 on Occasions With Sexual Stimulation- Change From Baseline
Description: Mean change: mean change at each visit minus mean at baseline. Percent of "Yes" responses to SEP Question 2 based on occasions (= sexual stimulation): 100*(number of occasions where SEP Question 3 [Did your erection last long enough for you to have successful intercourse?] = Yes) / (number of occasions where SEP Question 3 was answered Yes or No)
Time Frame: Week 2, Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 102
per-patient percentage
  Question 3 (Week 2) N=102 | 56.96 (38.93)
  Question 3 (Week 4) N=100 | 70.78 (35.46)
  Question 3 (Week 6) N=97 | 71.23 (35.79)
  Question 3 (Week 6 LOCF) N=102 | 72.15 (35.41)
  Question 3 (Week 6 Endpoint) N=100 | 71.60 (35.55)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 56.96, 95% CI [49.31 to 64.60], Standard Deviation 38.93
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 70.78, 95% CI [63.74 to 77.81], Standard Deviation 35.46
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 71.23, 95% CI [64.02 to 78.45], Standard Deviation 35.79
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 72.15, 95% CI [65.20 to 79.11], Standard Deviation 35.41
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 71.60, 95% CI [64.54 to 78.65], Standard Deviation 35.55

25. Secondary Outcome: Mean Per-Patient Percentage of 'Yes' Responses to Sexual Encounter Profile (SEP) Question 3 Based on Occasions With Sexual Stimulation- Change From Week 2
Description: Mean change: mean change at each visit minus mean at Week 2. Percent of "Yes" responses to SEP Question 2 based on occasions (= sexual stimulation): 100*(number of occasions where SEP Question 3 [Did your erection last long enough for you to have successful intercourse?] = Yes) / (number of occasions where SEP Question 3 was answered Yes or No)
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
per-patient percentage
  Question 3 (Week 4) N=110 | 13.56 (30.89)
  Question 3 (Week 6) N=107 | 14.25 (31.31)
  Question 3 (Week 6 LOCF) N=112 | 14.51 (31.77)
  Question 3 (Week 6 Endpoint) N=110 | 14.77 (32.00)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 13.56, 95% CI [7.72 to 19.40], Standard Deviation 30.89
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 14.25, 95% CI [8.25 to 20.25], Standard Deviation 31.31
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 14.51, 95% CI [8.56 to 20.46], Standard Deviation 31.77
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 14.77, 95% CI [8.72 to 20.82], Standard Deviation 32.00

26. Secondary Outcome: Mean Per-Patient Percentage of 'Yes' Responses to Sexual Encounter Profile (SEP) Question 4 Based on Occasions With Sexual Stimulation- Change From Baseline
Description: Mean change: mean change at each visit minus mean at baseline. Percent of "Yes" responses to SEP Question 4 based on occasions (= sexual stimulation): 100*(number of occasions where SEP Question 4 ["Were you satisfied with the hardness of your erection?"] = "Yes") / (number of occasions where SEP Question 4 was answered "Yes" or "No").
Time Frame: Week 2, Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 102
per-patient percentage
  Question 4 (Week 2) N=102 | 58.58 (41.24)
  Question 4 (Week 4) N=100 | 76.29 (37.21)
  Question 4(Week 6) N=97 | 77.69 (37.26)
  Question 4 (Week 6 LOCF) N=102 | 78.79 (36.65)
  Question 4 (Week 6 Endpoint) N=100 | 78.36 (36.89)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 58.58, 95% CI [50.48 to 66.68], Standard Deviation 41.24
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 76.29, 95% CI [68.90 to 83.67], Standard Deviation 37.21
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 77.69, 95% CI [70.18 to 85.21], Standard Deviation 37.26
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 78.79, 95% CI [71.59 to 85.99], Standard Deviation 36.65
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 78.36, 95% CI [71.04 to 85.68], Standard Deviation 36.89

27. Secondary Outcome: Mean Per-Patient Percentage of 'Yes' Responses to Sexual Encounter Profile (SEP) Question 4 Based on Occasions With Sexual Stimulation- Change From Week 2
Description: Mean change: mean change at each visit minus mean at Week 2. Percent of "Yes" responses to SEP Question 4 based on occasions (= sexual stimulation): 100*(number of occasions where SEP Question 4 ["Were you satisfied with the hardness of your erection?"] = "Yes") / (number of occasions where SEP Question 4 was answered "Yes" or "No").
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
per-patient percentage
  Question 4 (Week 4) N=110 | 17.90 (36.63)
  Question 4 (Week 6) N=107 | 19.50 (36.84)
  Question 4 (Week 6 LOCF) N=112 | 19.52 (36.99)
  Question 4 (Week 6 Endpoint) N=110 | 19.88 (37.23)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 17.90, 95% CI [10.98 to 24.83], Standard Deviation 36.63
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 19.50, 95% CI [12.44 to 26.56], Standard Deviation 36.84
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 19.52, 95% CI [12.59 to 26.45], Standard Deviation 36.99
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 19.88, 95% CI [12.84 to 26.91], Standard Deviation 37.23

28. Secondary Outcome: Mean Per-Patient Percentage of 'Yes' Responses to Sexual Encounter Profile (SEP) Question 5 Based on Occasions With Sexual Stimulation- Change From Baseline
Description: Mean change: mean change at each visit minus mean at baseline. Percent of "Yes" responses to SEP Question 5 based on occasions (= sexual stimulation): 100*(number of occasions where SEP Question 5 ["Were you satisfied with this sexual encounter?"] = "Yes") / (number of occasions where SEP Question 5 was answered "Yes" or "No")
Time Frame: Week 2, Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 102
per-patient percentage
  Question 5 (Week 2) N=101 | 57.34 (42.60)
  Question 5 (Week 4) N=100 | 70.72 (40.30)
  Question 5 (Week 6) N=97 | 70.63 (40.78)
  Question 5 (Week 6 LOCF) N=102 | 72.07 (40.27)
  Question 5 (Week 6 Endpoint) N=100 | 71.51 (40.48)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 57.34, 95% CI [48.93 to 65.75], Standard Deviation 42.60
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 70.72, 95% CI [62.72 to 78.71], Standard Deviation 40.30
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 70.63, 95% CI [62.41 to 78.85], Standard Deviation 40.78
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 72.07, 95% CI [64.16 to 79.98], Standard Deviation 40.27
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 71.51, 95% CI [63.48 to 79.55], Standard Deviation 40.48

29. Secondary Outcome: Mean Per-Patient Percentage of 'Yes' Responses to Sexual Encounter Profile (SEP) Question 5 Based on Occasions With Sexual Stimulation- Change From Week 2
Description: Mean change: mean change at each visit minus mean at Week 2. Percent of "Yes" responses to SEP Question 5 based on occasions (= sexual stimulation): 100*(number of occasions where SEP Question 5 ["Were you satisfied with this sexual encounter?"] = "Yes") / (number of occasions where SEP Question 5 was answered "Yes" or "No")
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 111
per-patient percentage
  Question 5 (Week 4) N=109 | 13.10 (29.11)
  Question 5 (Week 6) N=106 | 14.11 (32.53)
  Question 5 (Week 6 LOCF) N=111 | 13.47 (31.92)
  Question 5 (Week 6 Endpoint) N=109 | 13.72 (32.16)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 13.10, 95% CI [7.58 to 18.63], Standard Deviation 29.11
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 14.11, 95% CI [7.84 to 20.37], Standard Deviation 32.53
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 13.47, 95% CI [7.47 to 19.47], Standard Deviation 31.92
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 13.72, 95% CI [7.61 to 19.82], Standard Deviation 32.16

30. Secondary Outcome: Mean Per-Patient Percentage of 'Yes' Responses to Sexual Encounter Profile (SEP) Question 3 (Q3) Based on Attempts With Sexual Stimulation- Change From Baseline
Description: Mean change: mean change at each visit minus mean at baseline. Percent of "Yes" responses to SEP Q3 based on attempts with sexual stimulation (SS): 100* (number of attempts with SS where SEP Q3 [Did your erection last long enough for you to have successful intercourse?] = Yes)/(number of attempts with SS where SEP Q3 was answered Yes or No)
Time Frame: Week 2, Week 4, and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 102
per-patient percentage
  Week 2 (N=102) | 56.96 (38.93)
  Week 4 (N=100) | 70.78 (35.46)
  Week 6 (N=97) | 71.23 (35.79)
  Week 6 LOCF (N=102) | 72.15 (35.41)
  Week 6 Endpoint (N=100) | 71.60 (35.55)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus Baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 56.96, 95% CI [49.31 to 64.60], Standard Deviation 38.93
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 70.78, 95% CI [63.74 to 77.81], Standard Deviation 35.46
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 71.23, 95% CI [64.02 to 78.45], Standard Deviation 35.79
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 72.15, 95% CI [65.20 to 79.11], Standard Deviation 35.41
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 71.60, 95% CI [64.54 to 78.65], Standard Deviation 35.55

31. Secondary Outcome: Mean Per-Patient Percentage of 'Yes' Responses to Sexual Encounter Profile (SEP) Question 3 (Q3) Based on Attempts With Sexual Stimulation- Change From Week 2
Description: Mean change: mean change at each visit minus mean at Week 2. Percent of "Yes" responses to SEP Q3 based on attempts with sexual stimulation (SS): 100* (number of attempts with SS where SEP Q3 [Did your erection last long enough for you to have successful intercourse?] = Yes)/(number of attempts with SS where SEP Q3 was answered Yes or No)
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
per-patient percentage
  Week 4 (N=110) | 13.56 (30.89)
  Week 6 (N=107) | 14.25 (31.31)
  Week 6 LOCF (N=112) | 14.51 (31.77)
  Week 6 Endpoint (N=110) | 14.77 (32.00)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 13.56, 95% CI [7.72 to 19.40], Standard Deviation 30.89
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 14.25, 95% CI [8.25 to 20.25], Standard Deviation 31.31
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 14.51, 95% CI [8.56 to 20.46], Standard Deviation 31.77
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 14.77, 95% CI [8.72 to 20.82], Standard Deviation 32.00

32. Secondary Outcome: Mean Per-Patient Percentage of Grade 1 Events in Erection Hardness Grading Scale (EHGS) Based on Occasions With Sexual Stimulation- Change From Baseline
Description: Mean change: mean change at each visit minus mean at baseline. Percent of Grade 1 (1=increase in size, but not hard) erection hardness based on occasions: 100*(number of occasions where Erection Hardness Scale Answer 1)/(number of occasions where Erection Hardness Scale was answered)
Time Frame: Week 2, Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 103
per-patient percentage
  Grade 1 (Week 2) N=103 | -12.58 (37.77)
  Grade 1 (Week 4) N=101 | -20.55 (35.04)
  Grade 1 (Week 6) N=98 | -22.53 (36.64)
  Grade 1 (Week 6 LOCF) N=103 | -21.44 (36.06)
  Grade 1 (Week 6 Endpoint) N=101 | -21.86 (36.29)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus baseline; Test type: Superiority or Other; p = 0.0010, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -12.58, 95% CI [-19.96 to -5.20], Standard Deviation 37.77
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -20.55, 95% CI [-27.47 to -13.64], Standard Deviation 35.04
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -22.53, 95% CI [-29.88 to -15.18], Standard Deviation 36.64
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -21.44, 95% CI [-28.49 to -14.39], Standard Deviation 36.06
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -21.86, 95% CI [-29.03 to -14.70], Standard Deviation 36.29

33. Secondary Outcome: Mean Per-Patient Percentage of Grade 1 Events in Erection Hardness Grading Scale (EHGS) Based on Occasions With Sexual Stimulation- Change From Week 2
Description: Mean change: mean change at each visit minus mean at Week 2. Percent of Grade 1 (1=increase in size, but not hard) erection hardness based on occasions: 100*(number of occasions where Erection Hardness Scale Answer 1)/(number of occasions where Erection Hardness Scale was answered)
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
per-patient percentage
  Grade 1 (Week 4) N=110 | -6.79 (22.58)
  Grade 1 (Week 6) N=107 | -6.85 (23.02)
  Grade 1 (Week 6 LOCF) N=112 | -7.43 (24.20)
  Grade 1 (Week 6 Endpoint) N=110 | -7.57 (24.40)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p = 0.0021, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -6.79, 95% CI [-11.06 to -2.52], Standard Deviation 22.58
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p = 0.0027, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -6.85, 95% CI [-11.26 to -2.43], Standard Deviation 23.02
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p = 0.0015, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -7.43, 95% CI [-11.97 to -2.90], Standard Deviation 24.20
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p = 0.0015, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -7.57, 95% CI [-12.18 to -2.96], Standard Deviation 24.40

34. Secondary Outcome: Mean Per-Patient Percentage of Grade 2 Events in Erection Hardness Grading Scale (EHGS) Based on Occasions With Sexual Stimulation - Change From Baseline
Description: Mean change: mean change at each visit minus mean at baseline. Percent of Grade 2 (2= hard, but not hard enough for penetration) erection hardness based on occasions: 100*(number of occasions where Erection Hardness Scale Answer 2)/(number of occasions where Erection Hardness Scale was answered)
Time Frame: Week 2, Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 103
Per-patient percentage
  Grade 2 (Week 2) N=103 | -9.87 (34.44)
  Grade 2 (Week 4) N=101 | -11.74 (32.80)
  Grade 2 (Week 6) N=98 | -12.78 (33.56)
  Grade 2 (Week 6 LOCF) N=103 | -13.13 (33.94)
  Grade 2 (Week 6 Endpoint) N=101 | -12.40 (33.13)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus baseline; Test type: Superiority or Other; p = 0.0045, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -9.87, 95% CI [-16.60 to -3.14], Standard Deviation 34.44
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -11.74, 95% CI [-18.22 to -5.27], Standard Deviation 32.80
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -12.78, 95% CI [-19.51 to -6.05], Standard Deviation 33.56
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -13.13, 95% CI [-19.76 to -6.50], Standard Deviation 33.94
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -12.40, 95% CI [-18.94 to -5.86], Standard Deviation 33.13

35. Secondary Outcome: Mean Per-Patient Percentage of Grade 2 Events in Erection Hardness Grading Scale (EHGS) Based on Occasions With Sexual Stimulation - Change From Week 2
Description: Mean change: mean change at each visit minus mean at Week 2. Percent of Grade 2 (2= hard, but not hard enough for penetration) erection hardness based on occasions: 100*(number of occasions where Erection Hardness Scale Answer 2)/(number of occasions where Erection Hardness Scale was answered)
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
per-patient percentage
  Grade 2 (Week 4) N=110 | -2.39 (22.00)
  Grade 2 (Week 6) N=107 | -1.91 (20.73)
  Grade 2 (Week 6 LOCF) N=112 | -2.71 (22.28)
  Grade 2 (Week 6 Endpoint) N=110 | -2.76 (22.48)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p = 0.2567, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -2.39, 95% CI [-6.55 to 1.77], Standard Deviation 22.00
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p = 0.3435, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -1.91, 95% CI [-5.88 to 2.07], Standard Deviation 20.73
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p = 0.2000, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -2.71, 95% CI [-6.89 to 1.46], Standard Deviation 22.28
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p = 0.2000, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -2.76, 95% CI [-7.01 to 1.48], Standard Deviation 22.48

36. Secondary Outcome: Mean Per-Patient Percentage of Grade 3 Events in Erection Hardness Grading Scale (EHGS) Based on Occasions With Sexual Stimulation - Change From Baseline
Description: Mean change: mean change at each visit minus mean at baseline. Percent of Grade 3 (3= hard enough for penetration [but not completely hard]) erection hardness based on occasions: 100*(number of occasions where Erection Hardness Scale Answer 3)/(number of occasions where Erection Hardness Scale was answered)
Time Frame: Week 2, Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 103
per-patient percentage
  Grade 3 (Week 2) N=103 | -10.82 (56.75)
  Grade 3 (Week 4) N=101 | -29.16 (59.81)
  Grade 3 (Week 6) N=98 | -30.79 (60.90)
  Grade 3 (Week 6 LOCF) N=103 | -30.27 (61.70)
  Grade 3 (Week 6 Endpoint) N=101 | -30.87 (60.54)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus baseline; Test type: Superiority or Other; p = 0.0558, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -10.82, 95% CI [-21.91 to 0.27], Standard Deviation 56.75
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -29.16, 95% CI [-40.96 to -17.35], Standard Deviation 59.81
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -30.79, 95% CI [-43.00 to -18.58], Standard Deviation 60.90
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -30.27, 95% CI [-42.33 to -18.21], Standard Deviation 61.70
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -30.87, 95% CI [-42.82 to -18.92], Standard Deviation 60.54

37. Secondary Outcome: Mean Per-Patient Percentage of Grade 3 Events in Erection Hardness Grading Scale (EHGS) Based on Occasions With Sexual Stimulation - Change From Week 2
Description: Mean change: mean change at each visit minus mean at Week 2. Percent of Grade 3 (3= hard enough for penetration [but not completely hard]) erection hardness based on occasions: 100*(number of occasions where Erection Hardness Scale Answer 3)/(number of occasions where Erection Hardness Scale was answered)
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
per-patient percentage
  Grade 1 (Week 4) N=110 | -18.36 (46.03)
  Grade 1 (Week 6) N=107 | -22.16 (45.24)
  Grade 1 (Week 6 LOCF) N=112 | -20.28 (45.86)
  Grade 1 (Week 6 Endpoint) N=110 | -20.65 (46.20)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Median Difference (Net) = -18.36, 95% CI [-27.05 to -9.66], Standard Deviation 46.03
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -22.16, 95% CI [-30.84 to -13.49], Standard Deviation 45.24
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -20.28, 95% CI [-28.87 to -11.69], Standard Deviation 45.86
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = -20.65, 95% CI [-29.38 to -11.92], Standard Deviation 46.20

38. Secondary Outcome: Mean Per-Patient Percentage of Grade 4 Events in Erection Hardness Grading Scale (EHGS) Based on Occasions With Sexual Stimulation - Change From Baseline
Description: Mean change: mean change at each visit minus mean at baseline. Percent of Grade 4 (4= completely hard) erection hardness based on occasions: 100*(number of occasions where Erection Hardness Scale Answer 4)/(number of occasions where Erection Hardness Scale was answered)
Time Frame: Week 2, Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 103
per-patient percentage
  Grade 4 (Week 2) N=103 | 33.27 (41.43)
  Grade 4 (Week 4) N=101 | 61.45 (44.77)
  Grade 4 (Week 6) N=98 | 66.10 (45.15)
  Grade 4 (Week 6 LOCF) N=103 | 64.84 (45.70)
  Grade 4 (Week 6 Endpoint) N=101 | 65.13 (45.56)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 33.27, 95% CI [25.17 to 41.36], Standard Deviation 41.43
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 61.45, 95% CI [52.61 to 70.29], Standard Deviation 44.77
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 66.10, 95% CI [57.05 to 75.16], Standard Deviation 45.15
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 64.84, 95% CI [55.91 to 73.77], Standard Deviation 45.70
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 65.13, 95% CI [56.14 to 74.12], Standard Deviation 45.56

39. Secondary Outcome: Mean Per-Patient Percentage of Grade 4 Events in Erection Hardness Grading Scale (EHGS) Based on Occasions With Sexual Stimulation - Change From Week 2
Description: Mean change: mean change at each visit minus mean at Week 2. Percent of Grade 4 (4= completely hard) erection hardness based on occasions: 100*(number of occasions where Erection Hardness Scale Answer 4)/(number of occasions where Erection Hardness Scale was answered)
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 112
per-patient percentage
  Grade 4 (Week 4) N=110 | 27.53 (40.19)
  Grade 4 (Week 6) N=107 | 30.92 (41.90)
  Grade 4 (Week 6 LOCF) N=112 | 30.43 (41.88)
  Grade 4 (Week 6 Endpoint) N=110 | 30.98 (42.06)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 27.53, 95% CI [19.94 to 35.13], Standard Deviation 40.19
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 30.92, 95% CI [22.89 to 38.95], Standard Deviation 41.90
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 30.43, 95% CI [22.59 to 38.27], Standard Deviation 41.88
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 30.98, 95% CI [23.04 to 38.93], Standard Deviation 42.06

40. Secondary Outcome: Mean Per-Patient Percentage of Grade 3 or 4 Events in Erection Hardness Grading Scale (EHGS) Based on Occasions With Sexual Stimulation - Change From Baseline
Description: Mean change: mean change at each visit minus mean at baseline. Percent of Grade 3 (hard enough for penetration [but not completely hard]) or 4 (completely hard) erection hardness based on occasions: 100*(number of occasions where Erection Hardness Scale Answer 3 or 4)/ (number of occasions where Erection Hardness Scale was answered)
Time Frame: Week 2, Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 103
per-patient percentage
  Grade 3 or 4 (Week 2) N=103 | 22.45 (46.10)
  Grade 3 or 4 (Week 4) N=101 | 32.30 (42.15)
  Grade 3 or 4 (Week 6) N=98 | 35.31 (43.52)
  Grade 3 or 4 (Week 6 LOCF) N=103 | 34.57 (43.48)
  Grade 3 or 4 (Week 6 Endpoint) N=101 | 34.26 (43.29)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 2 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 22.45, 95% CI [13.44 to 31.46], Standard Deviation 46.10
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 4 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 32.30, 95% CI [23.97 to 40.62], Standard Deviation 42.15
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 35.31, 95% CI [26.59 to 44.04], Standard Deviation 43.52
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 34.57, 95% CI [26.07 to 43.07], Standard Deviation 43.48
Statistical Analysis 5: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 34.26, 95% CI [25.72 to 42.81], Standard Deviation 43.29

41. Secondary Outcome: Mean Per-Patient Percentage of Grade 3 or 4 Events in Erection Hardness Grading Scale (EHGS) Based on Occasions With Sexual Stimulation - Change From Week 2
Description: Mean change: mean change at each visit minus mean at Week 2. Percent of Grade 3 (hard enough for penetration [but not completely hard]) or 4 (completely hard) erection hardness based on occasions: 100*(number of occasions where Erection Hardness Scale Answer 3 or 4)/ (number of occasions where Erection Hardness Scale was answered)
Time Frame: Week 4 and Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per-patient percentage
Arm/Group | Open Label Sildenafil Citrate
Number analyzed (Participants) | 110
per-patient percentage
  Grade 3 or 4 (Week 4) N=110 | 9.18 (29.45)
  Grade 3 or 4 (Week 6) N=107 | 8.75 (29.26)
  Grade 3 or 4 (Week 6 LOCF ) N=112 | 10.15 (31.11)
  Grade 3 or 4 (Week 6 Endpoint ) N=110 | 10.33 (31.36)
Statistical Analysis 1: Comparison: Open Label Sildenafil Citrate; Week 4 minus Week 2; Test type: Superiority or Other; p = 0.0014, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 9.18, 95% CI [3.61 to 14.74], Standard Deviation 29.45
Statistical Analysis 2: Comparison: Open Label Sildenafil Citrate; Week 6 minus Week 2; Test type: Superiority or Other; p = 0.0025, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 8.75, 95% CI [3.15 to 14.36], Standard Deviation 29.26
Statistical Analysis 3: Comparison: Open Label Sildenafil Citrate; Week 6 LOCF minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 10.15, 95% CI [4.32 to 15.97], Standard Deviation 31.11
Statistical Analysis 4: Comparison: Open Label Sildenafil Citrate; Week 6 Endpoint minus Week 2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value not adjusted for multiple comparisons. Threshold for statistical significance p<0.05; single sample t-test; Mean Difference (Net) = 10.33, 95% CI [4.41 to 16.26], Standard Deviation 31.36

ADVERSE EVENTS:
Arm/Group | Open Label Sildenafil Citrate
Serious Adverse Events (participants affected / at risk) | 0/117
Other Adverse Events (participants affected / at risk) | 33
OTHER ADVERSE EVENTS (reported when occurring in more than 1.70% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Open Label Sildenafil Citrate
Headache (Nervous system disorders) | 18/117
Hot Flush (Vascular disorders) | 10/117
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3/117
Flushing (Vascular disorders) | 3/117
Gastritis (Gastrointestinal disorders) | 3/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.